CLINICAL TRIAL: NCT00633282
Title: Role of Pioglitazone and Berberine in Treatment of Non-alcoholic Fatty Liver Disease(NAFLD) Patients With Impaired Glucose Regulation or Type 2 Diabetes Mellitus
Brief Title: Role of Pioglitazone and Berberine in Treatment of Non-Alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xin Gao (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Sponsor-Investigator, Xin Gao, MD. and Professor, Vice-President of Zhongshan Hospital, Director of Department of Endocrinology & Metabolism of Zhongshan Hospital Fudan University, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07JC14011
Record Dates: First submitted 2008-03-03; First posted 2008-03-12 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Nonalcoholic Fatty Liver Disease; Pioglitazone; Berberine; Impaired Glucose Metabolism
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Exercise; Pioglitazone; Thiazolidinediones; Berberine; Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lifestyle intervention (Experimental): Life style intervention including aerobic exercise and reducing energy intake(-500kcal) without drug
  Interventions: Behavioral: Life style intervention
- Life style intervention, pioglitazone (Experimental): Life style intervention with pioglitazone 15mg qd for 16 weeks
  Interventions: Behavioral: Life style intervention; Drug: pioglitazone
- Life style intervention, berberine (Experimental): Life style intervention with berberine 0.5g tid for 16 weeks
  Interventions: Behavioral: Life style intervention; Drug: berberine

INTERVENTIONS:
Behavioral: Life style intervention — calorie limited diet: to subtract 500 kcal from daily mean calorie intake when entering the treatment
  activity: medium intensity aerobic exercise for more than 150 min per week with heart rate around 50-70% of the maximal heart rate; or higher-intensity aerobic exercise for more than 90min per week with heart rate around 70% of the maximal heart rate
  Other Names: calorie limited diet; aerobic exercise
Drug: pioglitazone — pioglitazone tablet,15mg qd ,30 minutes before breakfast,for 16 weeks
  Other Names: Actlns; PPAR agonist; Thiazolidinediones; insulin sensitizer
  Arms: Life style intervention, pioglitazone
Drug: berberine — berberine tablet 0.5g tid,30 minutes before each meal,for 16 weeks
  Other Names: traditional Chinese medicine; herb
  Arms: Life style intervention, berberine

SUMMARY:
The purpose of this study is to evaluate the effects and safety of pioglitazone and berberine on the basis of lifestyle intervention to non-alcoholic fatty liver disease patients with impaired glucose regulation or type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Sedentary lifestyle and poor dietary choices are leading to a weight gain epidemic and increasing the risk for developing nonalcoholic fatty liver disease (NAFLD). NAFLD is a group of diseases with too much fat in liver in the absence of excess alcohol consumption. NAFLD encompasses a histological spectrum ranging from simple hepatic steatosis to nonalcoholic steatohepatitis (NASH), advanced fibrosis, and cirrhosis. NAFLD is estimated to affect 25% of the worldwide population[1] and 15.35% of adults in shanghai urban area[2]. Epidemiological data showed that the fatty liver may predict, independent of other factors, the metabolic syndrome, type 2 diabetes, and cardiovascular disease. Therefore, we may prevent those diseases by treating NAFLD.Life style intervention including activity and reducing energy intake is recommended by health care providers for optimal health and is the most common prescribed therapy for individuals diagnosed with NAFLD.

TZDs are oral glucose-lowering medications used to treat type 2 diabetes that enhance insulin sensitivity. The strong relationship between insulin resistance and NAFLD suggests that insulin sensitizing therapies such as TZDs might be beneficial in the prevention or improvement in NAFLD.TZDs bind to the peroxisome proliferator-activated receptors (PPARs), in part, by facilitating enhanced TG storage by adipocytes, suppressing the ectopic storage of lipids into liver and skeletal muscle. In addition, TZDs appear to have anti-inflammatory properties, inhibiting adipocyte gene expression and reducing circulating levels of TNFα[3] and resistin[4], and increasing adiponectin concentrations[5]. Some researches demonstrated that pioglitazone(a TZD) significantly reduced liver fat content of NAFLD, and ameliorated biological parameters and liver histology of NASH[6]. However, there have not been similar data of treating chinese NAFLD with pioglitazone.

Berberine (BBR), a compound isolated from a Chinese herb was identified by Weijia [7] as a new cholesterol-lowering drug with a mechanism different from that of statin drugs. BBR elevates LDL receptor(LDLR) expression through a post-transcriptional mechanism that stabilizes the LDLR-mRNA. Considering the close relationship between NAFLD and lipid metabolism, we assume that BBR may be effective for NAFLD by improving lipid metabolism.

In order to evaluate these hypotheses, we plan to treat a group of NAFLD patients with impaired glucose regulation (IGR) or T2DM with pioglitazone or BBR in a randomized, open, controlled trial for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have an age range between 18 to 65 years (inclusive).
2. Patients with fatty liver confirmed by ultrasound.
3. Patients must meet the criteria for impaired glucose regulation or type 2 diabetes mellitus (FPG ≥ 5.6 mmol/L and/or a two hour glucose value ≥ 7.8 mmol/L).
4. Course of diabetic mellitus no more than 1 years
5. Diabetic patients have not received anti-diabetic drugs, including insulin, biguanides, sulfonylureas, thiazolidinediones, Alpha-glucosidase inhibitors, or glinides for 4 weeks before the time of enrollment
6. Patients have not received lipid-regulating drugs (statins, fibrates)for 4 weeks before the time of enrollment
7. Blood pressure < 160/100 mmHg,after receiving lifestyle therapy and effective anti-hypertensive drugs.
8. Patients must stopped other drugs medications for four weeks prior to entering the treatment period, such as: silybin, ursodeoxycholic acid, Polyene Phosphatidylcholine, vitamin E, some herbs with effect of regulating lipid and protecting liver function, etc.
9. Liver fat content(LFC) assessed by 1H MRS ≥ 13%(LFC was calculated by dividing the integral of the methylene groups in fatty acid chains of the hepatic triglycerides by the sum of methylene groups and water).

Exclusion Criteria:

1. Any causes of chronic liver disease other than NAFLD (such as - but not restricted to - alcohol or drug abuse, medication, chronic hepatitis B or C, autoimmune, etc.);
2. Patients with significantly impaired liver function: ALT or AST ≥ 2 times upper limit of normal;
3. HBsAg (+) and/or HCV-Ab (+);
4. Patients with type 1 diabetes mellitus or gestational diabetes or special type diabetes, and patients with BMI < 22 Kg/m2;
5. Course of diabetes more than 1 years;
6. Diabetics patients who have taken or are taking oral glucose-lowering drugs or insulin;
7. Diabetics patients with a HbA1c > 7.5% on initial visit;
8. Patients with severe diabetes complications (diabetes ketoacidosis, diabetes coma or with symptomatic of diabetes coma; dysfunction of nerve, retinopathy, dysfunction of kidney）;
9. Patients with serum creatinine ≥ 1.5 mg/dL (133 umol/L);
10. Patients with a history of clinically significant heart disease (myocardial infarct, heart failure, and or severe cardiac rhythm);
11. Complicating severe infection, within 6 months after operation, severe trauma;
12. Patients with excess alcohol consumption≥140g/week(male); ≥ 70g/week(female);
13. Patients have participated other clinical trials within 24 weeks;
14. Patients with a history of drug allergy to TZDs and berberine;
15. Patients wth gestation or possible gestation or lactation, or males or females who expecting gestation during clinical trial;
16. Mental diseases patients;
17. Those who refuse to sign informed consent;
18. Any other conditions, which, in the opinion of the investigators would impede competence or compliance or possibility of hindering completion of the study;
19. Patients with serum triglyceride ≥ 5.0 mmol/L;
20. Patients with thyroid disease, including hyperthyroidism or hypothyroidism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2008-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Improved metabolic parameters(glucose, lipid, liver enzymes, etc.) | 16 weeks
  improvement of the metabolic parameters, including serum glucose of OGTT, fasting glucose,2 hour glucose,area under the glucose curve and HbA1c,lipid profile（TC、TG、HDL-c、LDL-c、ApoA、ApoB、ApoE and Lpa），liver enzymes（ALT,AST,ALP,γ-GT）.

SECONDARY OUTCOMES:
liver fat content | 16 weeks
  improvement of liver fat content by 1H NMR spectroscopy
serum insulin | 16 weeks
  improvement of serum insulin including fasting insulin,2 hour insulin and area under insulin curve.
the ratio of withdrawing because of inefficiency | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xin GAO, MD, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - Endocrinology and Metabolism Department, Zhongshan Hospital, Fudan University,, Shanghai, Shanghai Municipality
  - Department of Endocrinology and Metabolism,Shanghai Clinical Center of Diabetes,Shanghai Institute of Diabetes,The sixth people's Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Department of Endocrinology and Metabolism,The Fifth People's Hospital，Fudan University, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Bedogni G, Miglioli L, Masutti F, Tiribelli C, Marchesini G, Bellentani S. Prevalence of and risk factors for nonalcoholic fatty liver disease: the Dionysos nutrition and liver study. Hepatology. 2005 Jul;42(1):44-52. doi: 10.1002/hep.20734. PMID 15895401
- [Background] Fan JG, Zhu J, Li XJ, Chen L, Li L, Dai F, Li F, Chen SY. Prevalence of and risk factors for fatty liver in a general population of Shanghai, China. J Hepatol. 2005 Sep;43(3):508-14. doi: 10.1016/j.jhep.2005.02.042. PMID 16006003
- [Background] Miyazaki Y, Mahankali A, Wajcberg E, Bajaj M, Mandarino LJ, DeFronzo RA. Effect of pioglitazone on circulating adipocytokine levels and insulin sensitivity in type 2 diabetic patients. J Clin Endocrinol Metab. 2004 Sep;89(9):4312-9. doi: 10.1210/jc.2004-0190. PMID 15356026
- [Background] Szapary PO, Bloedon LT, Samaha FF, Duffy D, Wolfe ML, Soffer D, Reilly MP, Chittams J, Rader DJ. Effects of pioglitazone on lipoproteins, inflammatory markers, and adipokines in nondiabetic patients with metabolic syndrome. Arterioscler Thromb Vasc Biol. 2006 Jan;26(1):182-8. doi: 10.1161/01.ATV.0000195790.24531.4f. Epub 2005 Nov 10. PMID 16284192
- [Background] Shadid S, Stehouwer CD, Jensen MD. Diet/Exercise versus pioglitazone: effects of insulin sensitization with decreasing or increasing fat mass on adipokines and inflammatory markers. J Clin Endocrinol Metab. 2006 Sep;91(9):3418-25. doi: 10.1210/jc.2006-0015. Epub 2006 Jun 27. PMID 16804048
- [Background] Yoneda M, Endo H, Nozaki Y, Tomimoto A, Fujisawa T, Fujita K, Yoneda K, Takahashi H, Saito S, Iwasaki T, Yamamoto S, Tsutsumi S, Aburatani H, Wada K, Hotta K, Nakajima A. Life style-related diseases of the digestive system: gene expression in nonalcoholic steatohepatitis patients and treatment strategies. J Pharmacol Sci. 2007 Oct;105(2):151-6. doi: 10.1254/jphs.fm0070063. Epub 2007 Oct 6. PMID 17928738
- [Background] Kong W, Wei J, Abidi P, Lin M, Inaba S, Li C, Wang Y, Wang Z, Si S, Pan H, Wang S, Wu J, Wang Y, Li Z, Liu J, Jiang JD. Berberine is a novel cholesterol-lowering drug working through a unique mechanism distinct from statins. Nat Med. 2004 Dec;10(12):1344-51. doi: 10.1038/nm1135. Epub 2004 Nov 7. PMID 15531889
- [Derived] Yan H, Wu W, Chang X, Xia M, Ma S, Wang L, Gao J. Gender differences in the efficacy of pioglitazone treatment in nonalcoholic fatty liver disease patients with abnormal glucose metabolism. Biol Sex Differ. 2021 Jan 4;12(1):1. doi: 10.1186/s13293-020-00344-1. PMID 33397443
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751
- [Derived] Chang X, Wang Z, Zhang J, Yan H, Bian H, Xia M, Lin H, Jiang J, Gao X. Lipid profiling of the therapeutic effects of berberine in patients with nonalcoholic fatty liver disease. J Transl Med. 2016 Sep 15;14:266. doi: 10.1186/s12967-016-0982-x. PMID 27629750
- [Derived] Yan HM, Xia MF, Wang Y, Chang XX, Yao XZ, Rao SX, Zeng MS, Tu YF, Feng R, Jia WP, Liu J, Deng W, Jiang JD, Gao X. Efficacy of Berberine in Patients with Non-Alcoholic Fatty Liver Disease. PLoS One. 2015 Aug 7;10(8):e0134172. doi: 10.1371/journal.pone.0134172. eCollection 2015. PMID 26252777